CLINICAL TRIAL: NCT03562078
Title: Tai Chi Quan Improving Blood Glucose, Blood Lipid, and Quality of Life in Patients With Type 2 Diabetes
Brief Title: Tai Chi Quan Improving Biochemistry and Quality of Life in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TaipeiCityH
Record Dates: First submitted 2018-04-18; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Tai Chi Quan; HbA1c; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Quan for Type 2 Diabetes (Experimental): diabetic patients care education and Tai Chi Quan training, including 10-minute warm-up, 40-minute Tai Chi lesson, and 10-minute cool-down exercise in the training, twice a week for 12 weeks.
  Interventions: Behavioral: Tai Chi Quan
- Control Group for Type 2 Diabetes (No Intervention): diabetic patients care education

INTERVENTIONS:
Behavioral: Tai Chi Quan — the first section of Yang style 108 form, including 10-minute warm-up, 40-minute training, and 10-minute cool-down exercise, twice a week
  Arms: Tai Chi Quan for Type 2 Diabetes

SUMMARY:
In this study, the hypothesis that the 12-week Tai Chi Quan training would have better control of blood sugar, biochemistry profile, and also better quality of life and activity of autonomic nerve system (ANS). The subjects were randomize assigned to either Tai Chi group or control group. The outcome measures before and after 12-week intervention include basic demographic characteristics, HbA1c, fasting blood glucose(FBG), triglycerides (TG), high and low density lipoprotein (HDL, LDL), creatinine(Cr), eGFR, GPT, ACR, quality of life, and activity of automatic nerve system.

DETAILED DESCRIPTION:
In this study, the hypothesis that the 12-week Tai Chi Quan training would have better control of blood sugar, biochemistry index, and also better quality of life and activity of automatic nerve system. In the study, type 2 diabetes mellitus(T2DM) patients will be recruited as subjects. The subjects were randomized to either Tai Chi group or control group. Tai Chi group would take Tai Chi Quan training for 1hr, twice a week for 12 weeks. There were 10-minute warm-up, 40-minute Tai Chi lesson, and 10-minute cool-down exercise in the training. In this study, the 1st section of Yang style 108 form is chosen for the experiment group. Both group were given diabetic patients care education and the exercise recording book for encouraging the daily exercise habits. The outcome measures before and after 12-week intervention include basic demographic characteristics, HbA1c, fasting blood glucose, triglycerides, high and low density lipid, creatinine, eGFR, GPT, ACR, quality of life, and activity of automatic nerve system.

ELIGIBILITY:
Inclusion Criteria:

* 40~80 years old
* Diagnosed type 2 diabetes mellitus, and without changing dietary pattern and medical treatment for blood glucose or blood lipid.
* Consciousness clear and is voluntary to attend the project and with the agreement.
* The functional movement ability is independent

Exclusion Criteria:

* Pregnant or plan to be pregnant in six months, and breast feeding.
* Severe complication in six months such as myocardial infarction, stroke, severe traumatic injury, major surgery. Other diseases evaluated by the doctor that are not suitable for the project.
* Evaluated that the compliance for the intervention is not appropriate.
* The blood glucose > 300mg/dl and unable to do vigorous exercise.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | change from Baseline to 12 weeks
  HbA1c

SECONDARY OUTCOMES:
fasting blood glucose | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
triglycerides | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
high and low density lipoprotein | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
creatinine | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
estimated Glomerular Filtration Rate (eGFR) | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
Glutamic-Pyruvic Transaminase (GPT) | change from Baseline to 12 weeks
  blood sample after 8-hour fasting
urine albumin/creatinine ratio (ACR) | change from Baseline to 12 weeks
  from urine sample
quality of life | change from Baseline to 12 weeks
  WHOQOL-BREF Taiwan
heart rate variability | change from Baseline to 12 weeks
  represent for balance of autonomic nervous system
low frequency (LF) | change from Baseline to 12 weeks
  Low frequency is the frequency domain analysis from heart rate variability, and is represent for sympathetic nervous system
high frequency (HF) | change from Baseline to 12 weeks
  High frequency is the frequency domain analysis from heart rate variability, and is represent for parasympathetic nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Jung Huang, Bachelor, Study Chair — Taipei City Hospital
Locations (1):
- Linsen Chinese Medicine and Kunming Branch, Taipei City Hospital, Taipei, Taiwan